CLINICAL TRIAL: NCT03403192
Title: A Comparison of Positional Stability: the EZ-blocker Versus Left Sided Double Lumen Tube in Adult Patients for Thoracic Surgery
Brief Title: EZ-blocker Versus Left Sided Double Lumen Tube in Adult Patients for Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00038220
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2019-06

CONDITIONS: Thoracic Injuries
Keywords: EZ Blocker; DLT; Double Lumen Tube; Thoracic Surgery
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Intervention Model Description: The objective of this study is to evaluate the positional stability and quality of lung isolation provided by the EZ-blocker compared to a DLT for both right and left sided thoracic surgery
Who Masked: Care Provider
Masking Description: The surgeon will be blinded to technique and queried as to the quality of isolation upon entry into the chest and this will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- EZ-Blocker in the left lung (Active Comparator): This arm will receive the EZ-Blocker in the left lung of their body, which functions as a bronchial blocker.
  Interventions: Device: EZ-Blocker
- EZ-Blocker in right lung (Active Comparator): This arm will receive the EZ-Blocker in the right lung of their body, which functions as a bronchial blocker.
  Interventions: Device: EZ-Blocker
- DLT in left lung (Active Comparator): This arm will receive the DLT in the left lung of their body, which functions as a bronchial blocker.
  Interventions: Device: DLT
- DLT in right lung (Active Comparator): This arm will receive the DLT in the right lung of their body, which functions as a bronchial blocker.
  Interventions: Device: DLT

INTERVENTIONS:
Device: EZ-Blocker — The EZ-Blocker essentially functions as a bronchial blocker with a 7-Fr shaft with two separate occlusive balloons coming off this shaft in a "Y" configuration designed to rest on the carina. Once anchored in place the operator can choose to inflate one of the two occlusive balloons to isolate one main stem bronchus or the other. According to the manufactures recommendations the EZ-blocker is placed through a Y-piece adaptor included with the blocker kit. A flexible fiberoptic bronchoscope (FFB) is placed in a separate limb of this Y-piece and this fed through along side the EZ-blocker to visualize and confirm placement of the of the BB. The balloon is then inflated typically under direct vision to occlude that bronchus thus isolating that lung hopefully achieving full lung isolation.
  Arms: EZ-Blocker in right lung; EZ-Blocker in the left lung
Device: DLT — A Double Lumen Tube (DLT) is made of two small-lumen endotracheal tubes of unequal length fixed side by side. The shorter tube ends in the trachea while the longer tube is placed in either the right or left bronchus to ventilate the right or left lung.
  Arms: DLT in left lung; DLT in right lung

SUMMARY:
The objective of this study is to evaluate the positional stability and quality of lung isolation provided by the EZ-blocker compared to a DLT for both right and left sided thoracic surgery.

An additional objective will be to assess time to placement of both devices and other significant clinical differences between these two approaches to placement of the bronchial blocker (BB) including airway injury and post-operatives sore throat, post-operative hoarseness, Additionally we would like to examine the preoperative high resolution CT imaging data to determine if there are anatomic landmarks that may potentially inform the appropriateness or inappropriateness of choosing an EZ-blocker or left sided DLT.

DETAILED DESCRIPTION:
One lung ventilation (OLV) is frequently used in thoracic surgery to promote surgical exposure and improve operative conditions. At this time, there are two different approaches to OLV in routine use in adult thoracic surgery. One approach is to use of a double lumen tube (DLT). The other approach is to use a bronchial blocker (BB). Currently there are several different types of bronchial BBs on the market.

The EZ-Blocker essentially functions as a bronchial blocker with a 7-Fr shaft with two separate occlusive balloons coming off this shaft in a "Y" configuration designed to rest on the carina. Once anchored in place the operator can choose to inflate one of the two occlusive balloons to isolate one main stem bronchus or the other.

A number of studies have been performed comparing BBs to DLTs looking at time and ease of placement, differences in quality of lung isolation, and incidence of sore throat, hoarseness, and other morbidity associated with placement. A recent meta-analysis published by Clayton-Smith et al found that BBs are associated with fewer airway injuries when compared to DLTs. They found the quality of isolation to be equivalent between BBs and DLTs. While quality of isolation over all may be comparable, it has been demonstrated in several studies that positional stability of bronchial blockers such as the Arndt or Cohen, is frequently inferior to that of a DLT.

At this time, there are a small number of trials looking at the use of the EZ-blocker in adult patients. In one study published in 2013 the EZ-blocker was compared to the Cohen Flex-Tip blocker. In this study they found that time to place the EZ-blocker was in fact shorter and that overall the number of repositioning required was less with the EZ-blocker. In 2013, a study was published by Mourisse et al which compared DLT to the EZ-blocker. In this study they found initial malposition of both devices to be fairly equivalent, and time to placement was longer with the EZ-blocker. They also found more tracheal and bronchial injuries in the DLT group, but importantly they found that positional stability was equivalent. In both of these studies however they did not design their studies to effectively differentiate between right and left sided procedures when quantifying the need for BB repositioning. Because the takeoff of the right upper lobe bronchus is sometimes adjacent to, or proximal to the carina, it can impede effective isolation with a BB. Therefore, claims of positional stability may rely heavily on the laterality of the procedure, with right sided isolation being significantly more labile than left sided especially with respect to isolation using a BB.

According to the manufactures recommendations the EZ-blocker is placed through a Y-piece adaptor included with the blocker kit. A flexible fiberoptic bronchoscope (FFB) is placed in a separate limb of this Y-piece and this fed through alongside the EZ-blocker to visualize and confirm placement of the BB. The balloon is then inflated typically under direct vision to occlude that bronchus thus isolating that lung hopefully achieving full lung isolation.

In conclusion then, the study team feels that the potential morbidity of a DLT in terms of the potential for airway injury when compared to a BB suggests that further exploration of the possibility of equivalent positional stability between these devices is necessary. The team also feels that it is necessary to delineate the impact of laterality on the effectiveness of one technique for isolation versus the other.

In addition to this if there is a difference in stability in cases where right sided isolation via the EZ-blocker fails in the setting of multiple repositions or out and out failure the team would like to examine the preoperative high resolution CT data to determine if there are anatomic measurement which could potentially inform the appropriateness or inappropriateness of choosing a DLT over an EZ-blocker.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 and 80 years of age scheduled for thoracoscopic surgery or thoracotomy requiring lung isolation
* Patient presenting as an outpatient for elective thoracic surgery
* In patients scheduled for thoracic surgery.

Exclusion Criteria:

* History of difficult airway/intubation
* Patients suspected to have a difficult airway.
* Morbid obesity BMI >39
* Pregnancy
* Emergency status of surgery
* Thoracic surgery requiring a right sided double lumen tube

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin N Morris, MD, Principal Investigator — Assistant Professor
Locations (1):
- Wake Forest Baptist Hospital, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Mungroop HE, Wai PT, Morei MN, Loef BG, Epema AH. Lung isolation with a new Y-shaped endobronchial blocking device, the EZ-Blocker. Br J Anaesth. 2010 Jan;104(1):119-20. doi: 10.1093/bja/aep353. No abstract available. PMID 20007802
- [Background] Dumans-Nizard V, Liu N, Laloe PA, Fischler M. A comparison of the deflecting-tip bronchial blocker with a wire-guided blocker or left-sided double-lumen tube. J Cardiothorac Vasc Anesth. 2009 Aug;23(4):501-5. doi: 10.1053/j.jvca.2009.02.002. Epub 2009 Apr 10. PMID 19362014
- [Background] Campos JH, Hallam EA, Van Natta T, Kernstine KH. Devices for lung isolation used by anesthesiologists with limited thoracic experience: comparison of double-lumen endotracheal tube, Univent torque control blocker, and Arndt wire-guided endobronchial blocker. Anesthesiology. 2006 Feb;104(2):261-6, discussion 5A. doi: 10.1097/00000542-200602000-00010. PMID 16436844
- [Background] Knoll H, Ziegeler S, Schreiber JU, Buchinger H, Bialas P, Semyonov K, Graeter T, Mencke T. Airway injuries after one-lung ventilation: a comparison between double-lumen tube and endobronchial blocker: a randomized, prospective, controlled trial. Anesthesiology. 2006 Sep;105(3):471-7. doi: 10.1097/00000542-200609000-00009. PMID 16931978
- [Background] Clayton-Smith A, Bennett K, Alston RP, Adams G, Brown G, Hawthorne T, Hu M, Sinclair A, Tan J. A Comparison of the Efficacy and Adverse Effects of Double-Lumen Endobronchial Tubes and Bronchial Blockers in Thoracic Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):955-66. doi: 10.1053/j.jvca.2014.11.017. Epub 2014 Dec 2. PMID 25753765
- [Background] Kus A, Hosten T, Gurkan Y, Gul Akgul A, Solak M, Toker K. A comparison of the EZ-Blocker with a Cohen Flex-Tip blocker for one-lung ventilation. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):896-9. doi: 10.1053/j.jvca.2013.02.006. Epub 2013 Aug 16. PMID 23958073
- [Background] Mourisse J, Liesveld J, Verhagen A, van Rooij G, van der Heide S, Schuurbiers-Siebers O, Van der Heijden E. Efficiency, efficacy, and safety of EZ-blocker compared with left-sided double-lumen tube for one-lung ventilation. Anesthesiology. 2013 Mar;118(3):550-61. doi: 10.1097/ALN.0b013e3182834f2d. PMID 23299364
- [Background] Piccioni F, Vecchi I, Spinelli E, Previtali P, Langer M. Extraluminal EZ-blocker Placement for One-lung Ventilation in Pediatric Thoracic Surgery. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):e71-3. doi: 10.1053/j.jvca.2015.05.200. Epub 2015 May 27. No abstract available. PMID 26342270
- [Background] Templeton TW, Downard MG, Simpson CR, Zeller KA, Templeton LB, Bryan YF. Bending the rules: a novel approach to placement and retrospective experience with the 5 French Arndt endobronchial blocker in children <2 years. Paediatr Anaesth. 2016 May;26(5):512-20. doi: 10.1111/pan.12882. Epub 2016 Mar 9. PMID 26956889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
Started | 41 | 40 | 40 | 42
Completed | 37 | 36 | 37 | 36
Not Completed | 4 | 4 | 3 | 6
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Unable to respond | 0 | 1 | 0 | 0
Not completed — Incomplete | 3 | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Double Lumen Tube (DLT) in Left Lung: This arm will receive the DLT in the left lung of their body, which functions as a bronchial blocker.
  DLT: A Double Lumen Tube (DLT) is made of two small-lumen endotracheal tubes of unequal length fixed side by side. The shorter tube ends in the trachea while the longer tube is placed in either the right or left bronchus to ventilate the right or left lung.
- Double Lumen Tube (DLT) in Right Lung: This arm will receive the DLT in the right lung of their body, which functions as a bronchial blocker.
  DLT: A Double Lumen Tube (DLT) is made of two small-lumen endotracheal tubes of unequal length fixed side by side. The shorter tube ends in the trachea while the longer tube is placed in either the right or left bronchus to ventilate the right or left lung.
- Total: Total of all reporting groups
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | Double Lumen Tube (DLT) in Left Lung | Double Lumen Tube (DLT) in Right Lung | Total
Number analyzed (Participants) | 41 | 40 | 40 | 42 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.5) | 65.3 (12.4) | 66.2 (12.9) | 60.6 (11.7) | 63.5 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 15 | 22 | 76
  Male | 21 | 21 | 25 | 20 | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 40 | 40 | 42 | 163
Weight [Mean (Standard Deviation); unit: kilograms] | 81.0 (17.1) | 77.0 (17.7) | 82.9 (16.4) | 82.0 (20.0) | 80.7 (17.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (4.8) | 26.5 (5.0) | 28.3 (4.79) | 28.5 (5.6) | 27.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Double Lumen Tube (DLT) or Bronchial Blocker (BB) Replacements
Description: Positional stability of lung isolation by measuring number of replacements due to device moving too deep or too shallow (proximal) within the lung.
Time Frame: End of surgical procedure
Measure: Number; unit: Number of replacements
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
Number analyzed (Participants) | 41 | 40 | 40 | 42
Number of replacements | 13 | 14 | 14 | 13

2. Secondary Outcome: Time it Takes to Place for Double Lumen Tube (DLT) and EZ
Description: Time of placement for both devices
Time Frame: End of surgical procedure
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
Number analyzed (Participants) | 41 | 40 | 40 | 42
Minutes | 3.2 [2.7 to 4.5] | 3.3 [2.5 to 4.9] | 2.0 [1.5 to 3.9] | 2.6 [1.3 to 3.8]

3. Secondary Outcome: Quality of Lung Isolation Between Devices
Description: Measured at 1 hour intervals during operation on a scale of 1-3 with 1 being Excellent, 2 being Fair, and 3 being Poor.
Time Frame: End of surgical procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
Number analyzed (Participants) | 41 | 40 | 40 | 42
score on a scale | 2.76 (0.39) | 2.70 (0.48) | 2.92 (0.26) | 2.83 (0.37)

4. Secondary Outcome: Side Effects of Devices
Description: Sore throat/hoarseness postoperatively on a scale of 0-100 with 0 being No Sore Throat and 100 being Worst Sore Throat Imaginable.
Time Frame: 2 days post operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
Number analyzed (Participants) | 41 | 40 | 40 | 42
score on a scale | 0 [0 to 5] | 3 [0 to 13] | 5 [0 to 12] | 0 [0 to 7]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | EZ-Blocker in the Left Lung | EZ-Blocker in Right Lung | DLT in Left Lung | DLT in Right Lung
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03403192/Prot_SAP_003.pdf
  • Informed Consent Form (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03403192/ICF_000.pdf